CLINICAL TRIAL: NCT04325061
Title: Efficacy of Dexamethasone Treatment for Patients With ARDS Caused by COVID-19
Acronym: DEXA-COVID19
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Li Ka Shing Knowledge Institute (Unknown); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Jesus Villar, Senior scientist, Dr. Negrin University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001278-31
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Acute Respiratory Distress Syndrome Caused by COVID-19
Keywords: ARDS; COVID-19; multiple system organ failure
MeSH Terms: conditions — COVID-19; Multiple Organ Failure | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled, open-label trial involving mechanically ventilated adult patients with ARDS caused by confirmed COVID-19 infection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients will be treated with standard intensive care
- Dexamethasone (Active Comparator): Standard intensive care plus dexamethasone
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone (20 mg/iv/daily/from Day 1 of randomization during 5 days, followed by 10 mg/iv/daily from Day 6 to 10 of randomization
  Other Names: dexamethasone Indukern
  Arms: Dexamethasone

SUMMARY:
Background: There are no proven therapies specific for Covid-19. The full spectrum of Covid-19 ranges from asymptomatic disease to mild respiratory tract illness to severe pneumonia, acute respiratory distress syndrome (ARDS), multiorgan failure, and death. The efficacy of corticosteroids in viral ARDS remains controversial.

Methods: This is an internationally (Spain, Canada, China, USA) designed multicenter, randomized, controlled, open-label clinical trial testing dexamethasone in mechanically ventilated adult patients with established moderate-to-severe ARDS caused by confirmed Covid-19 infection, admitted in a network of Spanish ICUs. Eligible patients will be randomly assigned to receive either dexamethasone plus standard intensive care, or standard intensive care alone. Patients in the dexamethasone group will receive an intravenous dose of 20 mg once daily from day 1 to day 5, followed by 10 mg once daily from day 6 to day 10. The primary outcome is 60-day mortality. The secondary outcome is the number of ventilator-free days at 28 days. All analyses will be done according to the intention-to-treat principle.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is a catastrophic illness of multifactorial etiology characterized by a diffuse, severe inflammatory process of the lung leading to acute hypoxemic respiratory failure requiring mechanical ventilation (MV). Pulmonary infections are the leading causes of ARDS. Clinical and experimental research has established a strong association between dysregulated systemic and pulmonary inflammation and progression or delayed resolution of ARDS.

The COVID-19 pandemic is a critical moment for the world. Severe pneumonia is the main condition leading to ARDS requiring weeks of MV with high mortality (40-60%) in COVID-19 patients. There is no specific therapy for Covid-19, although patients are receiving drugs that are already approved for treating other diseases. There has been great interest in the role of corticosteroids to attenuate the pulmonary and systemic damage in ARDS patients because of their potent anti-inflammatory and antifibrotic properties. However, the efficacy of corticosteroids in viral ARDS remains controversial.

We justify the need of this study based on the positive results of a recent clinical trial by our group, showing that dexamethasone for 10 days was able to reduce the duration of mechanical ventilation (MV) and increase hospital survival in patients with ARDS from multiple causes (Villar J et al. Lancet Respir Med 2020). Dexamethasone has never been evaluated in viral ARDS in a randomized controlled fashion. Our goal in this study is to examine the effects of dexamethasone on hospital mortality and on ventilator-free days in patients with moderate-to-severe ARDS due to confirmed COVID-19 infection admitted into a network of Spanish intensive care units (ICUs).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older;
* positive reverse-transcriptase-polymerase-chain-reaction (RT-PCR) assay for COVID-19 in a respiratory tract sample;
* intubated and mechanically ventilated;
* acute onset of ARDS, as defined by Berlin criteria as moderate-to-severe ARDS,3 which includes: (i) having pneumonia or worsening respiratory symptoms, (ii) bilateral pulmonary infiltrates on chest imaging (x-ray or CT scan), (iii) absence of left atrial hypertension, pulmonary capillary wedge pressure <18 mmHg, or no clinical signs of left heart failure, and (iv) hypoxemia, as defined by a PaO2/FiO2 ratio of ≤200 mmHg on positive end-expiratory pressure (PEEP) of ≥5 cmH2O, regardless of FiO2.

Exclusion Criteria:

* Routine treatment with corticosteroids during the previous week irrespective of dose;
* Corticosteroid use within the previous 24 h of more than 20 mg of dexamethasone or equivalent;
* Patients with a known contraindication to corticosteroids;
* Decision by a physician that involvement in the trial is not in the patient's best interest;
* Pregnancy and breast-feeding;
* Participation in another therapeutic trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
60-day mortality | 60 days
  All-cause mortality at 60 days after enrollment

SECONDARY OUTCOMES:
Ventilator-free days | 28 days
  Number of ventilator-free days (VFDs) at Day 28 (defined as days being alive and free from mechanical ventilation at day 28 after enrollment, For patients ventilated 28 days or longer and for subjects who die, VFD is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, Principal Investigator — Hospital Universitario Dr. Negrin
Locations (24):
- Spain (24):
  - ICU, Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Dr. Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Department of Anesthesia, Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Intensive Care Unit, Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - AVI, Hospital Clinic, Barcelona
  - Cardiac ICU, Hospital Clinic, Barcelona
  - Department of Anesthesia, Hospital Clinic, Barcelona
  - Hepatic ICU, Hospital Clínic, Barcelona
  - UVIR, Hospital Clinic, Barcelona
  - Intensive Care Unit, Hospital General de Ciudad Real, Ciudad Real
  - Department of Anesthesia, Hospital Universitario La Princesa, Madrid
  - Intensive Care Unit, Hospital Universitario La Princesa, Madrid
  - Intensive Care Unit, Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Department of Anesthesia, Hospital Universitario La Paz, Madrid
  - Intensive Care Unit, Hospital Universitario La Paz, Madrid
  - Department of Anesthesia, Hospital Universitario Virgen de Arrixaca, Murcia
  - Intensive Care Unit, Hospital Universitario Virgen de la Arrixaca, Murcia
  - Department of Anesthesia, Hospital Unversitario Montecelo, Pontevedra
  - Anesthesia, Hospital General Universitario de Valencia, Valencia
  - Department of Anesthesia, Hospital Clinico Universitario, Valencia
  - Intensive Care Unit, Hospital Clinico Universitario, Valencia
  - Department of Anesthesia, Hospital Clínico Universitario, Valladolid
  - Anesthesia, Hospital Universitario Río Hortega, Valladolid
  - Intensive Care Unit, Hospital Universitario Río Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Villar J, Belda J, Anon JM, Blanco J, Perez-Mendez L, Ferrando C, Martinez D, Soler JA, Ambros A, Munoz T, Rivas R, Corpas R, Diaz-Dominguez FJ, Soro M, Garcia-Bello MA, Fernandez RL, Kacmarek RM; DEXA-ARDS Network. Evaluating the efficacy of dexamethasone in the treatment of patients with persistent acute respiratory distress syndrome: study protocol for a randomized controlled trial. Trials. 2016 Jul 22;17:342. doi: 10.1186/s13063-016-1456-4. PMID 27449641
- [Result] Villar J, Ferrando C, Martinez D, Ambros A, Munoz T, Soler JA, Aguilar G, Alba F, Gonzalez-Higueras E, Conesa LA, Martin-Rodriguez C, Diaz-Dominguez FJ, Serna-Grande P, Rivas R, Ferreres J, Belda J, Capilla L, Tallet A, Anon JM, Fernandez RL, Gonzalez-Martin JM; dexamethasone in ARDS network. Dexamethasone treatment for the acute respiratory distress syndrome: a multicentre, randomised controlled trial. Lancet Respir Med. 2020 Mar;8(3):267-276. doi: 10.1016/S2213-2600(19)30417-5. Epub 2020 Feb 7. PMID 32043986
- [Derived] Villar J, Anon JM, Ferrando C, Aguilar G, Munoz T, Ferreres J, Ambros A, Aldecoa C, Suarez-Sipmann F, Thorpe KE, Juni P, Slutsky AS; DEXA-COVID19 Network. Efficacy of dexamethasone treatment for patients with the acute respiratory distress syndrome caused by COVID-19: study protocol for a randomized controlled superiority trial. Trials. 2020 Aug 16;21(1):717. doi: 10.1186/s13063-020-04643-1. PMID 32799933